CLINICAL TRIAL: NCT05022641
Title: Evaluating Impact of Near Infrared Autofluorescence (NIRAF) Detection for Identifying Parathyroid Glands During Parathyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Vanderbilt University (Other)
Responsible Party: Principal Investigator, Paul Gauger, Ambulatory Care Clinical Chief, William J Fry Professor of Surgery and Professor of Surgery, Medical School, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HUM00192089; 5R01CA212147-02 (NIH)
Record Dates: First submitted 2021-08-22; First posted 2021-08-26 (Actual); Results first posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Parathyroid Adenoma; Parathyroid Neoplasms; Parathyroid Cancer; Hypercalcemia; Primary Hyperparathyroidism
Keywords: Parathyroidectomy; Intraoperative Parathyroid Identification; Near Infrared Autofluorescence; Persistent Hyperparathyroidism; Persistent Hypercalcemia; Failed Parathyroidectomy; Repeat Parathyroidectomy
MeSH Terms: conditions — Parathyroid Neoplasms; Hypercalcemia; Hyperparathyroidism, Primary | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Masking Description: Only participants will be masked to the intervention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- PTeye (Experimental): The surgeon will use the PTeye as an intraoperative tool to identify if a suspect tissue is a parathyroid or not, during the parathyroid surgery.
  Interventions: Device: PTeye
- Standard of Care (Other): The surgeon will rely solely on her/his surgical experience in identifying the parathyroid glands during the operations.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: PTeye — The surgeon will first take 5 baseline NIRAF measurements on the thyroid gland (or neck muscle, if thyroid is absent) using the disposable sterile fiber probe that is connected to the PTeye console (see Figure 1), as per device functionality requirements.
  Arms: PTeye
Other: Standard of Care — The surgeon will rely solely on her/his surgical experience in identifying the parathyroid glands during the operations.
  Arms: Standard of Care

SUMMARY:
This study will see if the use of near infrared autofluorescence (NIRAF) detection with an FDA-cleared device 'Parathyroid Eye (PTeye)' for identifying parathyroid glands (PGs) during parathyroidectomy (PTx) procedures is better than a surgeon's detection alone. It compares risk-benefits and outcomes in PTx patients where NIRAF detection with PTeye for parathyroid identification is either used or not used.

Parathyroidectomy - look at application of the technology to see if it assists during a parathyroidectomy.

DETAILED DESCRIPTION:
Prior to data collection, it was determined some additional outcome measures collected by the primary site would not be relevant to the trial for participating sites such as this site. Those outcomes were removed from this record.

ELIGIBILITY:
Inclusion Criteria:

* Primary hyperparathyroidism who will be undergoing parathyroid surgery
* Persistent primary hyperparathyroidism after having undergone a failed prior parathyroid surgery who will be undergoing repeat parathyroid surgery

Exclusion Criteria:

* Pregnant women (Those patients who could potentially will receive preoperative pregnancy testing, as is standard before general anesthesia. Any patients with positive pregnancy test results will not be included in the study.)
* Patients with concurrent parathyroid and thyroid disease that require total thyroidectomy
* Patients with secondary or tertiary hyperparathyroidism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Gauger, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cousart AG, Kiernan CM, Willmon PA, Thomas G, Wang TS, Gauger PG, Duh QY, Underwood HJ, Jackson A, Patel A, Mahadevan-Jansen A, Solorzano CC. Near-Infrared Autofluorescence for Parathyroid Detection During Endocrine Neck Surgery: A Randomized Clinical Trial. JAMA Surg. 2025 Sep 1;160(9):936-944. doi: 10.1001/jamasurg.2025.2233. PMID 40668552

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PTeye | Standard of Care
Started | 81 | 79
Completed (Participants were considered to have completed the trial if data was collected from them for the primary outcome measure.) | 81 | 79
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PTeye | Standard of Care | Total
Number analyzed (Participants) | 81 | 79 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (15.2) | 61.1 (15.5) | 61.2 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 65 | 124
  Male | 22 | 14 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 81 | 78 | 159
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 76 | 69 | 145
  Black | 3 | 6 | 9
  Asian | 1 | 3 | 4
  Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 81 | 79 | 160
Final Diagnosis [Count of Participants; unit: Participants] — Diagnosis was determined after undergoing procedure.
  Participants
    Primary sporadic hyperparathyroidism | 78 | 77 | 155
    Recurrent/persistent hyperparathyroidism | 3 | 0 | 3
    Other | 0 | 2 | 2
Preoperative PTH (pg/mL) [Mean (Standard Deviation); unit: pg/mL] | 125.9 (78) | 124.1 (66.4) | 125 (72.3)
Preoperative calcium (pg/dL) [Mean (Standard Deviation); unit: pg/dL] | 11.5 (4.4) | 10.8 (0.6) | 11.2 (3.2)
Preoperative vitamin D (mcg) [Mean (Standard Deviation); unit: mcg] | 37.7 (16) | 35.8 (15.2) | 36.8 (15.6)

OUTCOME MEASURES:

1. Primary Outcome: Average Number of Parathyroid Glands Identified
Description: Average number of parathyroid glands identified between the Experimental Group: Glands identified with naked eye + NIRAF vs. the Control Group: Glands identified with naked eye.
Time Frame: Measured within the procedure, generally not more than 2 hours
Measure: Mean (95% Confidence Interval); unit: parathyroid glands per patient
Arm/Group | PTeye | Standard of Care
Number analyzed (Participants) | 81 | 79
parathyroid glands per patient | 2.7 [2.4 to 2.9] | 2.6 [2.3 to 2.8]
Statistical Analysis 1: Comparison: PTeye vs Standard of Care; Test type: Superiority; p = .6, t-test, 2 sided

2. Secondary Outcome: Parathyroid Hormone (PTH) Levels 5-14 Days After Surgery
Description: Parathyroid hormone (PTH) levels 5-14 days after surgery. Higher levels could indicate failure of operation. Low levels could indicate temporary or permanent parathyroid damage.
Time Frame: 5-14 days after surgery
Population: Not all participants returned for this lab assessment during the 5-14 day data collection period. As such, no data for these participants was collected.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PTeye | Standard of Care
Number analyzed (Participants) | 52 | 58
pg/mL | 23 (26.9) | 25.3 (23.4)
Statistical Analysis 1: Comparison: PTeye vs Standard of Care; Test type: Superiority; p = .65, t-test, 2 sided

3. Secondary Outcome: Appropriate Intraoperative Parathyroid Hormone Drop
Description: >50% drop from baseline at 10 minutes post-resection
Time Frame: baseline to 10 minutes
Population: Some participants' data was not collected by the surgeons during the baseline-to-10-minute time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | PTeye | Standard of Care
Number analyzed (Participants) | 80 | 75
Participants
  Yes | 45 | 56
  No | 35 | 19
Statistical Analysis 1: Comparison: PTeye vs Standard of Care; Test type: Superiority; p = .02, Chi-squared

4. Secondary Outcome: Duration of Surgery
Description: Surgery duration in minutes
Time Frame: Measured within the procedure, generally not more than 2 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | PTeye | Standard of Care
Number analyzed (Participants) | 81 | 79
minutes | 92.3 (40.2) | 88.8 (42.3)
Statistical Analysis 1: Comparison: PTeye vs Standard of Care; Test type: Superiority; p = 0.6, t-test, 2 sided

5. Secondary Outcome: Number of Nights Spent in the Hospital After Parathyroidectomy
Description: Number of nights spent for postoperative recovery in the hospital after the surgical procedure.
Time Frame: 0-72 hours after PTx procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | PTeye | Standard of Care
Number analyzed (Participants) | 81 | 79
Participants
  0 nights | 77 | 76
  1 night | 4 | 3

6. Secondary Outcome: Number of Frozen Sections
Description: Total number of frozen sections conducted for patients undergoing repeat surgery or bilateral neck explorations. Frozen sections were conducted to confirm that the parathyroid tissue for the targeted over-acting parathyroid was removed. Results reflect whether participants had a frozen section conducted.
Time Frame: Immediate
Measure: Count of Participants; unit: Participants
Arm/Group | PTeye | Standard of Care
Number analyzed (Participants) | 81 | 79
Participants
  0 frozen sections taken | 49 | 47
  1 or more frozen sections taken | 32 | 32
Statistical Analysis 1: Comparison: PTeye vs Standard of Care; Test type: Superiority; p = .6, Chi-squared

ADVERSE EVENTS:
Time Frame: Up to 6-months after surgery.
Arm/Group | PTeye | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/79
Other Adverse Events (participants affected / at risk) | 0/81 | 0/79

LIMITATIONS AND CAVEATS:
The relatively small sample size may miss rare events such as operative failure. Additionally, inter-variability amongst the two surgeons and their surgical approaches adds more complexity. Lastly, these findings may only be generalizable to higher volume centers with more experienced surgeons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-05): https://cdn.clinicaltrials.gov/large-docs/41/NCT05022641/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-05): https://cdn.clinicaltrials.gov/large-docs/41/NCT05022641/ICF_001.pdf